CLINICAL TRIAL: NCT06218823
Title: Comparative Effectiveness Trial of Tobacco Cessation Treatments Among Cancer Patients Who Smoke
Brief Title: Tobacco Treatment Comparison for Cancer Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1025; Protocol Version 2/13/2024 (Other: UW Madison); SMPH/MEDICINE/GEN INT MD (Other: UW Madison); 2P01CA180945-06 (NIH); UW23091 (Other: UWCCC)
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Smoking Cessation; Cancer
MeSH Terms: conditions — Smoking Cessation; Neoplasms | interventions — Tobacco Use Cessation Devices; Nicotine; Varenicline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low-Intensity Standard Smoking Cessation Treatment (Active Comparator): 2 weeks of nicotine patch therapy, 3 telephone counseling sessions, and information about quitline and National Cancer Institute text messaging support services (SmokefreeTXT)
  Interventions: Drug: Transdermal Nicotine Patch; Behavioral: Standard Telephone Counseling; Other: Mailed Information about Standard Care Resources
- High-Intensity, Cancer-Targeted Smoking Cessation Treatment (Experimental): 12 weeks of varenicline therapy, 7 counseling sessions targeted to cancer patients, and information about quitline and SmokefreeTXT services
  Interventions: Drug: Varenicline; Behavioral: Cancer-Targeted Telephone Counseling; Other: Mailed Information about Standard Care Resources

INTERVENTIONS:
Drug: Transdermal Nicotine Patch — a stop smoking aid, 21 milligrams(mg), 14mg, or 7mg of nicotine delivered over 24 hours
  Other Names: Nicotine Patch; NicoDerm CQ
  Arms: Low-Intensity Standard Smoking Cessation Treatment
Behavioral: Standard Telephone Counseling — 3 brief telephone-based smoking cessation counseling sessions
  Arms: Low-Intensity Standard Smoking Cessation Treatment
Drug: Varenicline — 12 weeks of an oral smoking cessation medication
  Other Names: apovarenicline
  Arms: High-Intensity, Cancer-Targeted Smoking Cessation Treatment
Behavioral: Cancer-Targeted Telephone Counseling — 7 telephone-based smoking cessation counseling sessions adapted for cancer patients
  Arms: High-Intensity, Cancer-Targeted Smoking Cessation Treatment
Other: Mailed Information about Standard Care Resources — Publicly funded treatment resources including the SmokefreeTXT program sponsored by the National Cancer Institute and the Wisconsin Tobacco Quit Line.

SUMMARY:
This pilot comparative effectiveness trial will compare two active smoking cessation treatments in terms of effectiveness, equity across patient subpopulations, and efficiency among adult patients diagnosed with cancer within the past 3 years. An enhanced treatment comprising 12 weeks of varenicline treatment and 7 smoking cessation coaching calls with a cancer focus will be compared against an active comparator modeled after standard quitline treatments (2 weeks of nicotine patch therapy with 3 phone coaching calls). Approximately 50 participants will be recruited to generate estimates of the effects, acceptability, costs, and equity of enhanced treatment (vs. standard treatment), with the primary outcome being abstinence from smoking 26 weeks after trying to quit.

DETAILED DESCRIPTION:
Primary Aim

1. To generate estimates of the size of the comparative effects of enhanced, cancer-specific smoking cessation treatment versus a generic standard care package similar to quitline care in terms of biochemically confirmed 7-day point prevalence abstinence (no smoking in the past 7 days) 26 weeks after a target quit date.

Exploratory Aims

1. To estimate differences in CET arms in exploratory outcomes including patient acceptability, completion, adherence, costs, and cost-effectiveness.
2. To estimate the extent to which treatment effects on abstinence and exploratory outcomes differ across patient subpopulations based on demographics (age, race, sex, ethnicity, socioeconomic disadvantage); nicotine dependence; and cancer site, stage, and treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Alive (per medical record)
* Diagnosed with cancer in the past 3 years
* Received care from a participating oncology clinic in the past year
* Has a current tobacco use status
* Does not have a preferred language other than English (missing language preference will be included).
* Valid address that is not a correctional facility or residential treatment/care facility.
* No flag for patient cognitive impairment, activated health care power of attorney, or other health care agent (e.g., legally authorized representative) in the EHR.

The following additional inclusion criteria must be met for inclusion in the CET

* Smoked combustible cigarettes in the past month.
* Able to speak and understand English.
* Willing to set a date to quit smoking in the next 60 days.
* Willing to receive smoking treatment information.
* Willing to complete study activities.

Exclusion Criteria:

* No current suicidal ideation.
* Suicide attempt in the past year.
* Currently receiving treatment for bipolar disorder, schizophrenia, schizoaffective disorder, or psychotic disorder.
* Incarceration.
* Unable to provide informed consent to treatment (i.e., cannot answer questions about study procedures or risks after hearing about the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E McCarthy, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate results from this research will be shared with the scientific community and our research collaborators. The findings from this research will also be shared upon request with study participants.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Data will only be shared under the auspices of an approved and executed Data Use Agreement, in accordance with university regulations.

REFERENCES:
- See also: UW Center for Tobacco Research and Intervention — https://ctri.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-Intensity Standard Smoking Cessation Treatment | High-Intensity, Cancer-Targeted Smoking Cessation Treatment
Started | 26 | 26
Completed | 23 | 24
Not Completed | 3 | 2
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Intensity Standard Smoking Cessation Treatment | High-Intensity, Cancer-Targeted Smoking Cessation Treatment | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (6.9) | 61.8 (8.3) | 64.0 (7.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 11 | 15 | 26
  Gender: Male | 14 | 10 | 24
  Gender: Other | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 24 | 23 | 47
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Biochemically Verified 7-day Point-prevalence Abstinence 26 Weeks After a Target Quit Date.
Description: This measure is confirmed by expired carbon monoxide and/or a cotinine urine or saliva sample test.
Time Frame: up to 30 weeks post target quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Intensity Standard Smoking Cessation Treatment | High-Intensity, Cancer-Targeted Smoking Cessation Treatment
Number analyzed (Participants) | 26 | 26
Participants | 2 | 7

2. Secondary Outcome: Self-reported 7-day Point-prevalence Abstinence 12 Weeks After a Target Quit Date.
Description: This measure is a self-report response at the 12 week telephone follow-up to the question "Have you smoked, even a puff, in the last 7 days?".
Time Frame: up to 13 weeks post target quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Intensity Standard Smoking Cessation Treatment | High-Intensity, Cancer-Targeted Smoking Cessation Treatment
Number analyzed (Participants) | 26 | 26
Participants | 6 | 9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline until 26 weeks.
Arm/Group | Low-Intensity Standard Smoking Cessation Treatment | High-Intensity, Cancer-Targeted Smoking Cessation Treatment
All-Cause Mortality (participants affected / at risk) | 3/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 8/26 | 6/26
Other Adverse Events (participants affected / at risk) | 4/26 | 8/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Intensity Standard Smoking Cessation Treatment (N=26) | High-Intensity, Cancer-Targeted Smoking Cessation Treatment (N=26)
Death (General disorders) | 3 (3) | 0 (0)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Hospitalization (Renal and urinary disorders) | 1 (1) | 1 (1)
Hospitalization (Cardiac disorders) | 1 (1) | 1 (1)
Hospitalization (General disorders) | 1 (2) | 3 (3)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Intensity Standard Smoking Cessation Treatment (N=26) | High-Intensity, Cancer-Targeted Smoking Cessation Treatment (N=26)
Nausea (Nervous system disorders) | 1 (1) | 3 (5)
Weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Vivid Dreams (Psychiatric disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT06218823/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT06218823/ICF_001.pdf